CLINICAL TRIAL: NCT02430844
Title: "Role of Biomarkers in Predicting Contrast-induced Acute Kidney Injury in Critically Ill Patients: a Prospective Observational Study"
Brief Title: Role of Biomarkers in Predicting Contrast-induced Acute Kidney Injury in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015-34-IMP-83
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; radiographic contrast; critically ill; biomarker
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Title: "Role of biomarkers in predicting contrast-induced acute kidney injury in critically ill patients: a prospective observational study"

Objective: To analyse the role of plasma and urinary biomarkers (Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1) in predicting contrast-induced acute kidney injury (CI-AKI) in critically ill patients.

Summary of the project:

Acute deterioration of renal function after intravenous administration of radiocontrast media, i.e. increase in serum creatinine concentration of more than 0.5 mg/dl or 25% above baseline within 48 hours, is referred to as contrast-induced kidney injury (CI-AKI). The increasing number of diagnostic procedures requiring radiographic contrast has parallel increase in the incidence of CI-AKI. CI-AKI is described as the third most common cause of new AKI in hospitalized patients. Occurrence of CI-AKI is reported up to 55% in high risk patients like presence pre-existing chronic renal dysfunction, diabetes, hypertension, chronic heart failure, advanced age, volume depletion, uses of concurrent nephrotoxic medication. These risk factors for CI-AKI are common in critically ill patients. Recently, different urinary and serum proteins have been intensively investigated as possible biomarkers for the early diagnosis of AKI, which includes Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1 (KIM 1). At present, there is scarcity of prospective study on CI-AKI and role of biomarkers in critically ill medical or medical-surgical mixed ICU patients.

The investigators plan to enroll about 100 ICU patients during 2 years, requiring computed tomography (CT) scans with parenteral administration of iodinated radiographic contrast for any diagnostic purposes as decided by the clinicians during the treatment of the patients. In this prospective observation study, the investigators want to analyse the role of plasma and urinary biomarkers in predicting CI-AKI in critically ill patients.

Key Words: acute kidney injury, radiographic contrast, critically ill, biomarker

DETAILED DESCRIPTION:
Rationale of the study supported by cited literature:

Role of biomarkers in AKI has been established in different clinical settings, to not only early diagnosis but also make prognosis. There are some studies in contrast-induced AKI, mainly in patients undergoing cardiac catheterization. Due to scarcity of prospective studies on this clinically important issue in critically ill patients, there is a need for this proposed study. The investigators will do study to analyse the role of plasma and urinary biomarkers (Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1) in predicting CI-AKI in critically ill patients

The relevance and expected outcome of the proposed study:

With this study, the investigators will be able to know that is there any predictive value of these biomarkers to predict CI-AKI in critically ill patients.

Preliminary work done so far:

No systematic study so far in critically ill medical-surgical ICU patients.

Definition of Contrast-induced acute kidney injury:

Contrast-induced acute kidney injury (CI-AKI) is defined as a rise in serum creatinine of ≥ 0.3 mg/dl from the baseline (before contrast exposure) value within 48 hours after administration of the radiographic contrast

Work plan methodology:

This is a prospective observational study to know role of biomarkers in CI-AKI in critically ill patients. Patients will be included from 2 intensive care units (ICU): 1. ICU of Department of Critical Care Medicine, and; 2. ICU of Department of Neurosurgery. All adult critically ill patients will be consider for inclusion in this study, who will require a contrast-enhanced CT scan of any organ system as decided by the treating clinician and also met study criteria as predefined. After getting written informed consent from the patient or close relatives to participate in this study, patients will be included in this study. There will be no intervention in this study. Treatment of patient will continue as per treating clinician. Transportation of patient for CT scanning will be accompanied by a senior resident and a staff nurse; and relevant monitoring of vitals will be done as per ICU protocol.

Sample collection: Sample will be collected after informed written consent. At baseline, before contrast exposure, 5 ml blood and 5 ml urine will be collected. Similar amount of each will be collected after 04 h, 24 h and 48 h of contrast exposure. Collected samples (plasma and urine) will be stored at temperature of -80 degree centigrade in deep freezer till analysis.

Data collection: Demographic and clinical characteristics of all ICU patients who fulfil inclusion criteria will be collected along with relevant laboratory tests done for patient management. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Dysfunction Assessment (SOFA) score will also be recorded. Contrast type and volume will be noted. Fluid balance in last 24 hours, uses of nephrotoxic drugs will also be noted.

Intervention: None. Outcome: The primary outcome measure will be development of contrast-induced acute kidney injury (CI-AKI), defined as a rise in plasma creatinine of ≥ 0.3 mg/dl from the baseline (before contrast exposure) value within 48 hours after administration of the radiographic contrast.

Laboratory methods: Samples will be analysed for plasma and urinary creatinine and studied biomarkers before contrast exposure as well as after 04 h, 24 h and 48 h of contrast exposure. Biomarker, Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1 (KIM 1) in plasma and urine, will be analysed by commercially available ELISA kits (RnD) as per manufacturer instructions. Urinary biomarker will be normalized as per urine creatinine values for each sample.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients who are > 18 years and having normal renal function, requiring radiographic contrast for diagnostic or interventional computed tomography procedure, will be considered for inclusion.

Exclusion Criteria:

* Age <18 years
* Known Chronic Kidney Disease
* Patient already on dialysis
* Presence of Acute Kidney Injury (increase in SCr by 50% or decrease in GFR by 25% within last 7 days)
* Recent exposure to radiographic contrast within 3 days of the study
* History of cardio/respiratory arrest during current illness
* Increase in serum creatinine levels of ≥ 0.3 mg/dl from the baseline during the previous 48 hours before contrast exposure.
* Known or suspected nephritic or nephrotic syndrome.
* A post-renal etiology of renal impairment
* Known allergy or hypersensitivity to radiographic contrast dye
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult critically ill patients having normal renal function will be consider for inclusion in this study, who will require a contrast-enhanced CT scan of any organ system as decided by the treating clinician and also met study criteria as predefined.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
To analyse the role of plasma and urinary biomarkers (Neutrophil Gelatinase-Associated Lipocalin (NGAL), Cystatin C and Kidney Injury Molecule-1) in predicting contrast-induced acute kidney injury (CI-AKI) in critically ill patients. | 48 Hours after contrast exposure
  Correlate levels of biomarkers in plasma and urine at different time interval in patients who develop contrast-induced acute kidney injury

OTHER OUTCOMES:
Incidence of contrast induced-acute kidney injury (CI-AKI) in critically ill patients | 48 Hours after contrast exposure
  Number of patients in whom Increase in serum creatinine >0.3 mg/dl within 48 hours after contrast media exposure

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS), Lucknow, Uttar Pradesh, India